CLINICAL TRIAL: NCT03388216
Title: A Phase I Study to Evaluate the Safety, Tolerance and Pharmacokinetics of the Anti-Shiga Toxin Hyperimmune Equine Immunoglobulin F(ab')2 Fragment (INM004) in Healthy Volunteers
Brief Title: Anti-Shiga Toxin Hyperimmune Equine Immunoglobulin F(ab')2 Fragment (INM004) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inmunova S.A. (Other)
Collaborators: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: CT-INM004-01
Record Dates: First submitted 2017-12-19; First posted 2018-01-02 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Stage I - Drug: INM004 Dose 1 (Experimental)
  Interventions: Biological: Drug: INM004 Dose 1
- Stage I - Placebo Dose 1 (Placebo Comparator)
  Interventions: Other: Placebo
- Stage I- Drug: INM004 Dose 2 (Experimental)
  Interventions: Biological: Drug: INM004 Dose 2
- Stage I- Placebo Dose 2 (Placebo Comparator)
  Interventions: Other: Placebo
- Stage II- Drug: INM004 Repeated Dose (Experimental)
  Interventions: Biological: Drug: INM004- Repeated dose
- Stage II- Placebo Repeated Dose (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Drug: INM004 Dose 1 — Stage I- Cohort I: (2mg/kg) administered at a single dose. The ratio is 3:1 (investigational product:placebo) -
  Arms: Stage I - Drug: INM004 Dose 1
Biological: Drug: INM004 Dose 2 — Stage I- Cohort II: Dose 2 (4mg/kg) administered at a single dose. The ratio is 3:1 (investigational product:placebo)
  Arms: Stage I- Drug: INM004 Dose 2
Biological: Drug: INM004- Repeated dose — Stage II: Either 3 doses of 2 mg/kg or 4 mg/kg will be administered every 24 hs. The ratio is 5:1 (investigational product : placebo).
  Arms: Stage II- Drug: INM004 Repeated Dose
Other: Placebo — A placebo infusion will be administered at the same infusion rate as the Drug arm
  Arms: Stage I - Placebo Dose 1; Stage I- Placebo Dose 2; Stage II- Placebo Repeated Dose

SUMMARY:
This is Prospective Randomized Placebo controlled Single Blind Phase I study to evaluate the safety, tolerance and pharmacokinetics of the anti-Shiga toxin hyperimmune equine immunoglobulin F(ab')2 fragment (INM004) in healthy volunteers.

DETAILED DESCRIPTION:
This is a study that will be conducted at a single site in Argentina to characterize the Pharmacokinetics (PK) profile, safety and tolerability of anti-Shiga toxin hyperimmune equine immunoglobulin F(ab')2 fragment (INM004) in 14 healthy subjects. This is a dose escalation study. Subjects will receive a single dose of an infusion of the biological product or placebo in Stage I where 2 cohorts will be assessed with 2 different doses of INM004. Subjects will receive a repeated dose (3 doses total, every 24 hs) of an infusion of the biological product or placebo in Stage II. The total duration of study participation is 4 weeks for each subject. Subjects will complete a follow-up visit at Day 30 after the dosing. Study duration is expected to last 6 months. The investigational product intent to use is for the prevention of the development of Hemolytic Uremic Syndrome (HUS) associated to Shigatoxin producing Escherichia coli (STEC).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index: between 19 and 27.
* Healthy subject, as determined by clinical exam, medical history and laboratory tests (chemistry, hematology and urine, pregnancy test if applicable) performed during the screening visit.
* Chest x-ray and electrocardiogram within normal ranges.

  -.Willing to participate and sign the informed consent.
* Women of child-bearing potential using at least two barrier birth control methods.
* Sexually active men using medically accepted birth control methods, such as condom with spermicide.

Exclusion Criteria:

* Known hypersensitivity to equine serum.
* Hypersensitivity to any of the components of the pharmaceutical preparation.
* History of severe allergic reactions to any type of antigen.
* History of mental illness.
* Participation in another clinical research study within 90 days6 months prior to the start of this study
* History of alcohol or drug abuse.
* History or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, hematological, neurological disease.
* Having received contrast substances for radiological studies of any kind in the two weeks prior to the start of the study.
* Receiving or having received any prescription drug within the two weeks prior to the start of the study, including oral contraceptives in women of child-bearing potential.
* Having received more than three doses of any over-the-counter medication during the week prior to the start of the study or any medication within two days prior to the hospitalization
* Having given blood within a period of under 2 months prior to the start of the study
* Documented infection with HIV, hepatitis B and/or hepatitis C.
* Pregnancy
* History of asthma, allergy, prior administration of equine serum (por example, anti-tetanus serum or anti-ophidic serum or anti-arachnid toxin serum) or allergic reaction due to contact or exposure to horses.
* History of vaccination within the month prior to the start of the study.
* Infectious disease requiring hospitalization within the month prior to the inclusion in the study.
* Having received a transfusion of blood products within three months prior to the inclusion in the study
* Having received any medication within 14 days prior to the inclusion in the study.
* Family relation or work relation to the personnel of the research group.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-12-16 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 4 weeks
Maximum Plasma Concentration [Cmax] | 4 weeks
Area Under the Curve [AUC] | 4 weeks
Elimination half-life (t½) | 4 weeks
Time of Maximum concentration observed (Tmax) | 4 weeks

SECONDARY OUTCOMES:
Number of participants with treatment-related hypersensitivity events as assessed by CTCAE v4.0 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Sanguineti, Ph.D, Study Director — Inmunova S.A.
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aire, Argentina

IPD SHARING:
Plan to Share IPD: Undecided